CLINICAL TRIAL: NCT01097369
Title: A Multicenter Registry Study of Anti-rasburicase Antibodies in Patients Retreated With Rasburicase (SR29142) in the Context of Relapsing Leukemia/Lymphoma Who Experienced Subsequent Hypersensitivity Reaction(s) or Loss of Uricolytic Activity: An Immuno-Monitoring Observational Study
Brief Title: Elitek (Rasburicase) Immuno-Monitoring Study
Status: Terminated | Type: Observational
Why Stopped: business decision due to low subject recruitment
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: RASBU_L_02990
Record Dates: First submitted 2010-03-31; First posted 2010-04-01 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Tumor Lysis Syndrome
MeSH Terms: conditions — Tumor Lysis Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Anti-rasburicase antibodies

SUMMARY:
Primary Objective:

To determine the incidence, titer and type of anti-rasburicase antibodies in the context of hypersensitivity reaction(s) or the loss of uricolytic activity occurring in patients with relapsed leukemia/lymphoma who have been re-treated with rasburicase and have experienced a hypersensitivity reaction or loss of uricolytic activity.

ELIGIBILITY:
Inclusion criteria:

1. Previous history of rasburicase exposure and history of administration of a repeat (2nd) series of rasburicase injections (in the context of supportive care for relapsing leukemia/lymphoma) and subsequent development of either a hypersensitivity reaction (HSR) or loss of uricolytic activity (defined as failure to achieve uric acid level of < or = 7.5 mg/dl measured 48 hours after the first rasburicase injection).

   1. A severe hypersensitivity reaction (NCI Grade 3, 4 or 5) is defined as:

      Allergic reaction; allergy; anaphylactic shock; bronchospasm; bullous skin eruption; dermatitis - exfoliative; drug hypersensitivity; dyspnea; hypotension; hypoxia; rash; rash - erythematous; rash - maculopapular, urticaria; pyrexia/fever; edema; chest discomfort; hypersensitivity (NOS); pharynx discomfort; hoarseness; pharyngeal erythema; pruritus; erythema; localized exfoliation; rash - papular; swelling ¿ face/facial; toxic skin eruption; hot flush; flushing; rash - macular; rash - pruritic; pruritus - allergic.
   2. Loss of uricolytic activity can be defined as:

      * uric acid levels > 7.5 mg/dl measured 48 hours after the first rasburicase injection¿, which is a time point coincident with administration of the third dose of rasburicase (within that second course of treatment with this agent).
2. Patients should have received at least 2 doses of rasburicase during the repeat (2nd) administration in the event of loss or uricolytic activity. At least 1 dose of rasburicase should be administered during the repeat (2nd) administration for diagnosis of HSR.

Exclusion criteria:

1. Concomitant treatment with human IV immunoglobulin (IVIG)
2. Concomitant treatment with TNF-alpha antagonists/inhibitors, i.e. adalimumab, infliximab, and etanercept
3. Concomitant treatment with Interferon-alpha (IFN-alpha)
4. Unwillingness or inability to comply with the requirements of the protocol.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients are selected as the clinical manifestations for study inclusion (hypersensitivity reaction or the loss of uricolytic activity) are recognized during clinically-indicated re-challenge with rasburicase.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2010-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Prevalence/frequency of presence of anti-rasburicase antibodies in eligible population. | Day 1, i.e. within 48 hours of identification /diagnosis of HSR (hypersensitivity reaction) or loss of uricolytic activity
Titer/type of anti-rasburicase antibodies in eligible population. | Day 1, i.e. within 48 hours of identification /diagnosis of HSR (hypersensitivity reaction) or loss of uricolytic activity

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (4):
- United States (4):
  - Investigational Site Number 3, Valhalla, New York
  - Investigational Site Number 4, Oklahoma City, Oklahoma
  - Investigational Site Number 2, Memphis, Tennessee
  - Investigational Site Number 1, Houston, Texas